CLINICAL TRIAL: NCT06867211
Title: Use of Ultrasonography for Measuring Achilles Tendon Thickness: a Novel Measurement Method
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Necip Gökhan Güner, Assistant Professor, MD, Sakarya University
Other Study IDs: 43012747-050.04-399468-15
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Achilles Tendon; Emergency Medicine; Ultrasonography
Keywords: achilles tendon; emergency medicine; ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Use of Ultrasonography for Measuring Achilles Tendon Thickness
  Interventions: Diagnostic Test: Use of Ultrasonography for Measuring Achilles Tendon Thickness

INTERVENTIONS:
Diagnostic Test: Use of Ultrasonography for Measuring Achilles Tendon Thickness — Achilles tendon ultrasonography was performed on healthy volunteers included in the study by an emergency physician trained in both basic and advanced ultrasonography techniques. Measurements were conducted using a Butterfly iQ (Butterfly Network, Inc., Guilford, CT) ultrasound device in B-mode with a musculoskeletal preset, using biplane imaging. For Achilles tendon measurement, the image depth was set to 2.0 cm. A linear probe was placed longitudinally and perpendicular to the tendon. The distal portion of the Achilles tendon and the calcaneus were visualized in the long axis, whereas the short axis was used to center the Achilles tendon on the screen for an optimal measurement view. The measurement site was determined as 2 cm proximal to the Achilles tendon insertion at the calcaneus. In biplane imaging, Achilles tendon thickness was measured in the long axis, whereas thickness, width, and cross-sectional area were measured in the short axis. Measurements were performed bilaterally

SUMMARY:
Background: Achilles tendon thickness has been associated with various diseases. Among imaging modalities, ultrasonography stands out because of its advantages in assessing Achilles tendon thickness. Previous studies typically recommend performing Achilles tendon ultrasonography with the patient in a prone position on an examination table. However, because it is not always possible or safe for each patient to assume the prone position, this study aimed to investigate the relationship between measurements obtained in the supine position and those obtained using the standard method.

Methods: A total of 180 healthy volunteers aged ≥18 years (70 female and 110 male; 360 Achilles tendons), with no history of disease or medication use, were included in the study. Achilles tendon measurements (thickness, width, and cross-sectional area) were obtained via ultrasonography in four different positions, including the standard method. The alternative methods included the supine position with the leg extended (Method 2), the supine position with the ankle resting on the opposite knee (Method 3), and the supine position with the leg held in the air at 90 degrees of hip and knee flexion (Method 4). Measurements were taken 2 cm distal from the Achilles tendon insertion on the calcaneus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged >18 years who agreed to participate in the study

Exclusion Criteria:

* Individuals with tenosynovitis, tendinitis, bursitis, tuberculous arthritis, rheumatoid arthritis, a history of Achilles tendon surgery, or tendon injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size for this study was calculated to include at least 180 volunteers, based on a moderate effect size, an error margin of 0.05, a power of 80%, and a correlation analysis approach.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
A novel ultrasonographic technique for achilles tendon thickness measurement | Baseline
  The primary outcome of this study was to provide a practical method for Achilles tendon measurement in emergency departments by addressing the disadvantages of the prone measurement technique proposed in previous studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharifaskari A, Goodarzi A, Davoody N, Kianmehr N, Sepyani A, Haghighi A. Sonographic assessment of Achilles tendon in patients with cutaneous psoriasis. Caspian J Intern Med. 2024 Spring;15(2):313-317. doi: 10.22088/cjim.15.2.313. PMID 38807726
- [Background] Tharwat S, Saleh M, Elrefaey R, Nassar MK, Nassar MK. Clinical and Ultrasonographic Characteristics of the Achilles Tendon in Hemodialysis Patients. Medicina (Kaunas). 2023 Dec 15;59(12):2181. doi: 10.3390/medicina59122181. PMID 38138284
- [Background] Silbernagel KG, Shelley K, Powell S, Varrecchia S. Extended field of view ultrasound imaging to evaluate Achilles tendon length and thickness: a reliability and validity study. Muscles Ligaments Tendons J. 2016 May 19;6(1):104-10. doi: 10.11138/mltj/2016.6.1.104. eCollection 2016 Jan-Mar. PMID 27331037
- [Background] Del Bano-Aledo ME, Martinez-Paya JJ, Rios-Diaz J, Mejias-Suarez S, Serrano-Carmona S, de Groot-Ferrando A. Ultrasound measures of tendon thickness: Intra-rater, Inter-rater and Inter-machine reliability. Muscles Ligaments Tendons J. 2017 May 10;7(1):192-199. doi: 10.11138/mltj/2017.7.1.192. eCollection 2017 Jan-Mar. PMID 28717629
- [Background] Yuzawa K, Yamakawa K, Tohno E, Seki M, Akisada M, Yanagi H, Okafuji T, Yamanouchi Y, Hattori N, Kawai K, et al. An ultrasonographic method for detection of Achilles tendon xanthomas in familial hypercholesterolemia. Atherosclerosis. 1989 Feb;75(2-3):211-8. doi: 10.1016/0021-9150(89)90178-0. PMID 2653326
- [Background] Steinmetz A, Schmitt W, Schuler P, Kleinsorge F, Schneider J, Kaffarnik H. Ultrasonography of achilles tendons in primary hypercholesterolemia. Comparison with computed tomography. Atherosclerosis. 1988 Dec;74(3):231-9. doi: 10.1016/0021-9150(88)90242-0. PMID 3071370
- [Background] Murugan A, Kanakaraju K, R M S, Sanjoy Mishra V. Achilles Tendon Softness and Thickness in Patients With Hypercholesterolemia. Cureus. 2022 Aug 24;14(8):e28340. doi: 10.7759/cureus.28340. eCollection 2022 Aug. PMID 36168354